CLINICAL TRIAL: NCT06907004
Title: Developing a Exercise Program for Patients Undergoing Hematopoietic Stem Cell Transplantation: An Action Research Approach.
Brief Title: Developing a Exercise Program for Patients Undergoing Hematopoietic Stem Cell Transplantation
Status: Completed | Type: Observational
Sponsor: Chimei Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 11111-006
Record Dates: First submitted 2025-03-19; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2023-02

CONDITIONS: Hematopoietic Stem Cell Transplantation
Keywords: Action research; Hematopoietic stem cell transplantation; Exercise program

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Background: Hematopoietic stem cell transplantation (HSCT) is a highly aggressive treatment, which is associated with numerous treatment-related side effects, such as fatigue and decreased functional activity. While recent studies have shown that physical exercise for patients undergoing HSCT is safe and feasible, and has a positive effect on the quality of life, fatigue, and lower limb muscle strength. However, there is no consensus regarding the intensity, type and frequency of exercise program, and few studies mention the patients' experience of exercise barriers and facilitators during HSCT. Therefore, the clinical implementation of exercise program is quite difficult.

Purpose: The purpose of this study is to develop a feasible exercise program for hospitalized patients undergoing hematopoietic stem cell transplantation.

Methods: Action Research is used to collect quantitative and qualitative data. Through the rolling revision of the exercise program during HSCT, finally develop a feasible exercise program.

Expected results: Developing a feasible exercise program for hospitalized patients undergoing hematopoietic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. First-time hematopoietic stem cell transplantation (HSCT) patients who are ambulatory, their primary caregivers, and physical therapists and nurses participating in the exercise intervention;
2. Age 20 years or older;
3. Capable of understanding and complying with the study objectives;
4. No psychiatric disorders or cognitive impairments.

Exclusion Criteria:

1. HSCT patients deemed unsuitable for exercise participation based on the attending physician's assessment;
2. HSCT patients at risk of fractures or confined to bed rest due to musculoskeletal conditions.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: First-time hematopoietic stem cell transplantation (HSCT) patients and their primary caregivers, and physical therapists and nurses at Chimei Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
Exercise adherence rate | approximately 4-6 weeks
  Definition: The percentage of prescribed exercise sessions completed by participants during the hematopoietic stem cell transplantation hospitalization period.
  Measurement Method:
  1. Numerator: Number of completed exercise sessions
  2. Denominator: Total number of prescribed exercise sessions
  3. Unit of Measure: Percentage (%)
Patient Satisfaction Score of the Exercise Program | approximately 4-6 weeks
  Definition: The mean score of a 7-item satisfaction questionnaire using a 5-point Likert scale to evaluate patient's satisfaction with the exercise program.
  Measurement Method:
  1. Tool: 7-item satisfaction questionnaire with 5-point Likert scale Scale Range: 1 (strongly disagree) to 5 (strongly agree)
  2. Total Score Calculation: Mean score of all 7 items
  3. Unit of Measure: Score on a scale (1-5)
  Questionnaire Items:
  1. Appropriateness of exercise timing
  2. Appropriateness of exercise intensity
  3. Appropriateness of exercise frequency
  4. Appropriateness of exercise type and difficulty level
  5. Achievement of exercise goals
  6. Satisfaction with personal performance
  7. Willingness to continue exercising
Exercise-Related Adverse Events Rate | approximately 4-6 weeks
  Definition: The percentage of exercise sessions with adverse events during the hematopoietic stem cell transplantation hospitalization period.
  Measurement Method:
  1. Numerator: Number of exercise sessions with adverse events
  2. Denominator: Total number of completed exercise sessions
  3. Unit of Measure: Percentage (%)

CONTACTS AND LOCATIONS:
Overall Officials: Min-Syuan Yen, Master's Degree, Principal Investigator — Chimei Medical Center
Locations (1):
- Chimei Medical Center, Tainan, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the following reasons:
  1. Privacy and confidentiality concerns - The study involves sensitive medical information from HSCT patients and personal experiences from healthcare providers.
  2. Ethical restrictions - The informed consent obtained from participants did not include permission for data sharing beyond the research team.
  3. Hospital policy compliance - The participating medical center's regulations restrict the sharing of patient-related data to protect patient privacy.
  4. Small sample size - With only 24 participants, sharing individual data might risk participant identification, even if anonymized.

REFERENCES:
- [Background] Morishita S, Nakano J, Fu JB, Tsuji T. Physical exercise is safe and feasible in thrombocytopenic patients with hematologic malignancies: a narrative review. Hematology. 2020 Dec;25(1):95-100. doi: 10.1080/16078454.2020.1730556. PMID 32075567
- [Background] Morishita S, Kaida K, Setogawa K, Kajihara K, Ishii S, Ikegame K, Kodama N, Ogawa H, Domen K. Safety and feasibility of physical therapy in cytopenic patients during allogeneic haematopoietic stem cell transplantation. Eur J Cancer Care (Engl). 2013 May;22(3):289-99. doi: 10.1111/ecc.12027. Epub 2012 Dec 18. PMID 23252444
- [Background] Mohammed J, Aljurf M, Althumayri A, Almansour M, Alghamdi A, Hamidieh AA, ElHaddad A, Othman TB, Bazarbachi A, Almohareb F, Alzahrani M, Alkindi SS, Alsharif F, Da'na W, Alhashmi H, Bekadja MA, Al-Shammari SH, El Quessar A, Satti TM, Aljohani N, Rasheed W, Ghavamzadeh A, Chaudhri N, Hashmi SK. Physical therapy pathway and protocol for patients undergoing hematopoietic stem cell transplantation: Recommendations from The Eastern Mediterranean Blood and Marrow Transplantation (EMBMT) Group. Hematol Oncol Stem Cell Ther. 2019 Sep;12(3):127-132. doi: 10.1016/j.hemonc.2018.12.003. Epub 2019 Jan 11. PMID 30653940
- [Background] Liang Y, Zhou M, Wang F, Wu Z. Exercise for physical fitness, fatigue and quality of life of patients undergoing hematopoietic stem cell transplantation: a meta-analysis of randomized controlled trials. Jpn J Clin Oncol. 2018 Dec 1;48(12):1046-1057. doi: 10.1093/jjco/hyy144. PMID 30277514
- [Background] Knols RH, de Bruin ED, Uebelhart D, Aufdemkampe G, Schanz U, Stenner-Liewen F, Hitz F, Taverna C, Aaronson NK. Effects of an outpatient physical exercise program on hematopoietic stem-cell transplantation recipients: a randomized clinical trial. Bone Marrow Transplant. 2011 Sep;46(9):1245-55. doi: 10.1038/bmt.2010.288. Epub 2010 Dec 6. PMID 21132025
- [Background] Campbell KL, Winters-Stone KM, Wiskemann J, May AM, Schwartz AL, Courneya KS, Zucker DS, Matthews CE, Ligibel JA, Gerber LH, Morris GS, Patel AV, Hue TF, Perna FM, Schmitz KH. Exercise Guidelines for Cancer Survivors: Consensus Statement from International Multidisciplinary Roundtable. Med Sci Sports Exerc. 2019 Nov;51(11):2375-2390. doi: 10.1249/MSS.0000000000002116. PMID 31626055
- See also: Physical Activity Guidelines for Taiwanese — https://www.hpa.gov.tw/Pages/EBook.aspx?nodeid=1411